CLINICAL TRIAL: NCT02626455
Title: A Phase III, Randomized, Double-blind, Controlled Multicenter Study of Intravenous PI3K Inhibitor Copanlisib in Combination With Standard Immunochemotherapy Versus Standard Immunochemotherapy in Patients With Relapsed Indolent Non-Hodgkin's Lymphoma (iNHL)
Brief Title: Study of Copanlisib in Combination With Standard Immunochemotherapy in Relapsed Indolent Non-Hodgkin's Lymphoma (iNHL)
Acronym: CHRONOS-4
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decided to terminate this study due to study did not meet the primary endpoint.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17833; 2015-001088-38 (EudraCT Number)
Record Dates: First submitted 2015-11-03; First posted 2015-12-10 (Estimated); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Clinical trial, Phase III; Phosphatidylinositol-3-kinase; Non-Hodgkin's lymphoma; Indolent B-cell non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — copanlisib; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Bendamustine Hydrochloride; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Copanlisib + R-B or R-CHOP / Arm 1 (Experimental): Combination of copanlisib with standard immunochemotherapy (rituximab and bendamustine) [R-B] or rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone [R-CHOP] (safety run-in and phase III)
  Interventions: Drug: Copanlisib (BAY80-6946); Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Bendamustine; Drug: Prednisone
- Placebo + R-B or R-CHOP / Arm 2 (Placebo Comparator): Combination of placebo and R-B or R-CHOP (phase III only)
  Interventions: Drug: Placebo; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Bendamustine; Drug: Prednisone

INTERVENTIONS:
Drug: Copanlisib (BAY80-6946) — Copanlisib is supplied as lyophilized preparation in a 6 mL injection vial. The total amount of copanlisib per vial is 60 mg. The solution for IV infusions is obtained after reconstitution with normal saline solution. For patients on R-B dosing of copanlisib will be administered on Days 1, 8 and 15 of each 28-day cycle. Copanlisib will be administered and then rituximab followed by bendamustine. For patients on R-CHOP dosing of copanlisib will be administered on Days 1 and 8 of each 21-day cycle. Treatment with copanlisib/placebo will be continued up to 12 months.
  Copanlisib will be administered before rituximab followed by cyclophosphamide, doxorubicin and vincristine infusions. Prednisone/prednisolone tablets to be taken for 5 days.
  Arms: Copanlisib + R-B or R-CHOP / Arm 1
Drug: Placebo — Placebo is supplied as lyophilized preparation in a 6 mL injection vial. The developed placebo lyophilisate is equivalent to the 60 mg copanlisib formulation, with regard to the composition of excipients and the instructions for reconstitution and dose preparation. Placebo dosing will be administered as per copanlisib described above. Applies to the phase III part of the study only.
  Arms: Placebo + R-B or R-CHOP / Arm 2
Drug: Rituximab — Rituximab is administered as an infusion at a dose of 375 mg/m2 body surface on Day 1 of each 28-day cycle for patients assigned to R-B and on Day 2 of each 21-day cycle for patients assigned to R-CHOP.
Drug: Cyclophosphamide — Cyclophosphamide is administered as an infusion at a dose of 750 mg/m2 body surface on Day 2 of each 21-day cycle for patients assigned to R-CHOP
Drug: Doxorubicin — Doxorubicin is administered as an infusion at a dose of 50 mg/m2 body surface on Day 2 of each 21-day cycle for patients assigned to R-CHOP
Drug: Vincristine — Vincristine is administered as an infusion at a dose of 1.4 mg/m2 body surface (maximum dose 2.0 mg) on Day 2 of each 21-day cycle for patients assigned to R-CHOP
Drug: Bendamustine — Bendamustine is administered as an infusion at a dose of 90 mg/m2 body surface on Day 1 and Day 2 for patients assigned to R-B
Drug: Prednisone — Prednisone is given as 100 mg tablets daily from Day 2 to Day 6 for patients assigned to R-CHOP

SUMMARY:
The purpose of this study is to assess whether copanlisib in combination with standard immunochemotherapy (rituximab in combination with bendamustine [R-B] and rituximab in combination with a 4 drug combination of cyclophosphamide, doxorubicin, vincristine and prednisone/prednisolone [R-CHOP]) is effective and safe, compared with placebo in combination with standard immunochemotherapy (R-B or R-CHOP) in patients with relapsed iNHL who have received at least one, but at most three, lines of treatment, including rituximab-based immunochemotherapy and alkylating agents.

DETAILED DESCRIPTION:
Patients should be in need of and fit for immunochemotherapy and should not be resistant to rituximab (resistance defined as lack of response or progression within 6 months of the last date of rituximab administration, including rituximab, and/or rituximab biosimilars, and/or anti-CD20 monoclonal antibody).

This study will be composed of two parts: Safety run-in and phase III part. The purpose of the safety run-in part of this study is to assess whether the drug being tested (copanlisib) in combination with standard immunochemotherapy (R-B or R-CHOP) is safe and at what dose level of the study drug (copanlisib - 45mg or 60 mg) patients are able to tolerate the study treatment combination. In addition to finding a safe and tolerable dose level for the phase III part of the study, efficacy will also be evaluated for patients that stay on the study treatment during the safety run-in. The phase III part of the study started with the determined recommended dose of copanlisib of 60 mg in combination with R-B. Combination treatment of copanlisib at the recommended/approved dose of 60 mg with R-B or R-CHOP was completed in April 2021.

A maximum of 24 patients will take part in the safety run-in part of this study. In the phase III part approximately 520 patients will be randomly assigned to blinded treatment arms of copanlisib plus R-B or R-CHOP or placebo plus R-B or R-CHOP. Combination therapy (copanlisib/placebo with R-B or R-CHOP) will be administered for a maximum of 6 cycles (C1-C6). Copanlisib/placebo (study drug) monotherapy will be administered from C7 onwards.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of B lymphocyte antigen CD20 positive iNHL with histological subtype limited to:

  * Follicular lymphoma G1-2-3a
  * Small lymphocytic lymphoma with absolute lymphocyte count <5x10E9/L at study entry
  * Lymphoplasmacytoid lymphoma / Waldenström macroglobulinemia (LPL / WM)
  * Marginal zone lymphoma (MZL) (splenic, nodal, or extra-nodal)
* Patients must have relapsed (recurrence after complete response or presented progression after partial response) or progressed after at least one but at most three prior lines of therapy, including rituximab, and/or rituximab biosimilars, and/or anti-CD20 monoclonal antibody (e.g. obinutuzumab) -based immunochemotherapy and alkylating agents (if given concomitantly is considered one line of therapy). A previous regimen is defined as one of the following: at least 2 months of single-agent therapy (less than 2 months of therapy with single agent rituximab, or rituximab biosimilars, or anti-CD20 monoclonal antibody can be considered a previous regimen in the case the patient responded to it); at least 2 consecutive cycles of polychemotherapy; autologous transplant; or radioimmunotherapy. Previous exposure to other PI3K Inhibitors (except copanlisib) is acceptable provided there is no resistance (resistance defined as no response (response defined as partial response [PR] or complete response [CR]) at any time during therapy, or progressive disease (PD) after any response (PR/CR) or after stable disease within 6 months from the end of the therapy with a PI3K inhibitor.
* Non-WM patients must have at least one bi-dimensionally measurable lesion (that has not been previously irradiated) according to the Lugano Classification. For patients with splenic MZL this requirement may be restricted to splenomegaly alone since that is usually the only manifestation of measurable disease.
* Patients affected by WM who do not have at least one bi-dimensionally measurable lesion in the baseline radiologic assessment must have measurable disease, defined as presence of immunoglobulin M (IgM) paraprotein with a minimum IgM level ≥ 2 x upper limit of normal and positive immunofixation test.
* Male or female patients ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Life expectancy of at least 3 months
* Availability of fresh tumor tissue and/or archival tumor tissue at Screening
* Adequate baseline laboratory values as assessed within 7 days before starting study treatment.
* Left ventricular ejection fraction ≥ 50%

Exclusion Criteria

* Histologically confirmed diagnosis of follicular lymphoma grade 3b or transformed disease, or chronic lymphocytic leukemia. In patients with clinical suspicion of transformed disease, a fresh biopsy is recommended.
* Rituximab, or rituximab biosimilars, or anti-CD20 monoclonal antibody (e.g. obinutuzumab) resistance at any line of therapy (resistance defined as lack of response, or progression within 6 months of the last date of rituximab, or rituximab biosimilars, or anti-CD20 monoclonal antibody administration, including maintenance with these drugs).
* HbA1c > 8.5% at screening
* History or concurrent condition of interstitial lung disease and/or severely impaired lung function (as judged by the investigator)
* Known lymphomatous involvement of the central nervous system
* Known history of human immunodeficiency virus (HIV) infection
* Hepatitis B (HBV) or hepatitis C (HCV) infection. Patients positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) will be eligible if they are negative for HBV-DNA, these patients should receive prophylactic antiviral therapy as per rituximab label. Patients positive for anti-HCV antibody will be eligible if they are negative for HCV-RNA.
* Cytomegalovirus (CMV) infection. Patients who are CMV PCR positive at baseline will not be eligible.CMV PCR test is considered positive if, the result can be interpreted as a CMV viremia according to local standard of care.
* Uncontrolled hypertension despite optimal medical management (per investigator´s assessment)
* Congestive heart failure > New York Heart Association (NYHA) class 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (201):
- United States (10):
  - Ironwood Physicians P.C. DBA Ironwood Cancer & Res. Ctr., Chandler, Arizona
  - Brian J. LeBerthon, MD, West Covina, California
  - SCL Health Research at St Joseph's Hospital Denver CO, Denver, Colorado
  - Lewis Hall Singletary Oncology Center, Thomasville, Georgia
  - Memorial Sloan Kettering Cancer Center- Bergen, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Cancer and Blood Specialists, Port Jefferson Station, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Oncology Consultants, Houston, Texas
  - Texas Oncology- McAllen, McAllen, Texas
- Australia (6):
  - Calvary Mater Hospital Newcastle, Waratah, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Ashford Cancer Centre Research Pty Ltd, Kurralta Park, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Eastern Health Integrated Renal Service, Box Hill
- Belgium (4):
  - Institut Jules Bordet/Jules Bordet Instituut, Brussels
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - CHU de Liège, Liège
- Brazil (10):
  - Centro Integrado de Oncologia de Curitiba, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericordia de Porto Alegre | Hospital Sao Francisco - Centro Medico Pesquisa Clinica Cardiologia, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre | Clinical Research Center - Surgery Research Center, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Oncológicas, Florianópolis, Santa Catarina
  - Faculdade de Ciencias Medicas-Universidade Estadual Campinas, Campinas, São Paulo
  - Centro Multidisciplinar de Estudos Clínicos EPP - Ltda., São Bernardo do Campo, São Paulo
  - IEP São Lucas, São Paulo, São Paulo
  - Instituto Nacional do Cancer Jose Alencar Gomes da Silva, Rio de Janeiro
  - Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo
  - Hospital Israelita Albert Einstein | Morumbi - Clinical Research Department, São Paulo
- Bulgaria (4):
  - UMHAT Sveti Georgi, Plovdiv
  - University Multiprofile Hosp. for Active Treat. Sveti Ivan, Sofia
  - SHATHD Spec. Hospi. for Active Treatm. of Haematol. Dis. EAD, Sofia
  - Multiprofile Hospital for Active Treatment Hristo Botev AD, Vratsa
- Canada (4):
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - Hopital de L'Enfant Jesus, Québec, Quebec
  - Centre Universitaire de Sante de l'Estrie, Sherbrooke, Quebec
- Chile (3):
  - Sociedad de Investigaciones Medicas Ltda, Temuco, Región de la Araucanía
  - Centro de Investigaciones Clínicas Vina del Mar Ltda., Viña del Mar, Región de Valparaíso
  - Instituto Nacional del Cáncer, Santiago
- China (18):
  - FuJian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Tumor Hospital of Hebei Province, Hebei, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - 1st Affiliated hospital of Soochow University, Suzhou, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The Affiliated Hospital of Qingdao University, Shandong, Shandong
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - The 1st Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Fifth Medical Center, General Hospital of the Chinese People, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Xinhua Hos Affiliated to SH Jiaotong Uni School of Medicine, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Tianjin Union Medicine Centre (People's Hospital of Tianjin), Tianjin
- Czechia (2):
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Kralovske Vinohrady, Prague
- Denmark (2):
  - Rigshospitalet - Hjertesygdomme, København Ø
  - Odense Universitetshospital - Hæmatologisk afdeling, Odense C
- Finland (4):
  - HUS, Meilahden sairaala, Helsinki
  - Oulun yliopistollinen sairaala, Oulu
  - Tampereen yliopistollinen sairaala, Tampere
  - Turun yliopistollinen keskussairaala, Turku
- France (12):
  - Centre Hospitalier Universitaire - Angers, Angers
  - Centre Hospitalier de la Durance - Avignon, Avignon
  - Centre Hospitalier Intercommunal de la Côte Basque-Bayonne, Bayonne
  - Centre Hospitalier Universite de Grenoble, Grenoble
  - Clinique Victor Hugo - Le Mans, Le Mans
  - Hôpital Dupuytren, Limoges
  - Hôpital Saint-Eloi, Montpellier
  - Hopital Hotel Dieu - Nantes, Nantes
  - Hôpital Saint Louis, Paris
  - Centre François Magendie - Pessac, Pessac
  - Hôpital de la Milétrie, Poitiers
  - Clinique Saint Anne, Strasbourg
- Germany (8):
  - Stauferklinikum Schwäbisch-Gmünd, Mutlangen, Baden-Wurttemberg
  - Haematologie-Onkologie im Zentrum MVZ GmbH, Augsburg, Bavaria
  - Klinikum der Universität München Grosshadern, München, Bavaria
  - Medizinische Hochschule Hannover (MHH), Hanover, Lower Saxony
  - Marienhospital Herne Universitätsklinik, Herne, North Rhine-Westphalia
  - Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia
  - Oncologianova GmbH, Recklinghausen, North Rhine-Westphalia
  - Med. Fakultät der Martin-Luther-Universität Halle-Wittenberg, Halle, Saxony-Anhalt
- Greece (5):
  - EVANGELISMOS General Hospital of Athens, Athens
  - General Hospital of Athens LAIKO, Athens
  - University General Hospital of Athens "ATTIKON", Chaïdári
  - Univ. General Hospital of Larissa, Larissa
  - University General Hospital of Patras, Pátrai
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Hungary (6):
  - Semmelweis University, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz, Nyíregyháza
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Komarom-Esztergom Varmegyei Szent Borbala Korhaz, Tatabánya
- Ireland (2):
  - Cork University Hospital, Cork
  - Mater Misericordiae University Hospital, Dublin
- Israel (4):
  - Rambam Health Corporation, Haifa
  - Hadassah Hebrew University Hospital Ein Kerem, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
  - Shamir Medical Center (Assaf Harofeh), Ẕerifin
- Italy (4):
  - IRCCS Ospedale Policlinico San Martino, Genoa, Liguria
  - Humanitas Mirasole S.p.A., Milan, Lombardy
  - IRCCS Fondazione Policlinico San Matteo, Pavia, Lombardy
  - A.O.U. Ospedali Riuniti "Umberto I - G.M.Lancisi - G.Salesi", Ancona, The Marches
- Japan (20):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - JCHO Kyushu Hospital, Kitakyushu, Fukuoka
  - Gunma University Hospital, Maebashi, Gunma
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Tenri Hospital, Tenri, Nara
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Aomori Prefectural Central Hospital, Aomori
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hiroshima Red Cross & Atomic-bomb Survivors Hospital, Hiroshima
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Kumamoto University Hospital, Kumamoto
  - Osaka Red Cross Hospital, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Yamagata University Hospital, Yamagata
- Mexico (5):
  - Hospital General de México SS, México, D. F., Mexico City
  - Centro de Investigación Clínica Chapultepec S.A. de C.V., Morelia, Michoacán
  - Hospital Universitario "José Eleuterio González", Monterrey, Nuevo León
  - Centro Especializado en Investigación Clínica S.C., Boca del Río, Veracruz
  - Centro de Atencion e Investigacion Clinica en Oncologia SCP, Mérida, Yucatán
- Poland (3):
  - Szpital Morski im. PCK, Gdynia
  - Pratia McM Kraków, Krakow
  - Wojew. Szpital Specjalistyczny im. M. Kopernika, Lodz
- Portugal (4):
  - Centro Clinico Academico Braga | Braga, Portugal, Braga
  - Centro Hospitalar Universitario do Porto, Porto
  - IPO Porto, Porto
  - Centro Hospitalar Vila Nova de Gaia e Espinho | Unit 1 - Clinical Research Center, Porto
- Romania (8):
  - Sp. Judetean de Urgenta Dr. Constantin Opris Baia Mare, Baia Mare
  - Sc Onco Card Srl, Brasov
  - Spitalul Clinic Colentina, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
- Russia (7):
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - Clinical Oncological Dispensary of Omsk Region, Omsk
  - Research Institute of Oncology, Rostov-on-Don
  - RSRI of Hematology and Transfusiology, Saint Petersburg
  - Oncology Dispensary #2, Sochi
  - Siberian State Medical University, Tomsk
  - Republican Clinical Oncology Dispensary, Ufa
- Singapore (3):
  - National University Hospital, Singapore
  - National Cancer Center Singapore, Singapore
  - Singapore General Hospital, Singapore
- Narodny onkologicky ustav, Bratislava, Slovakia
- South Africa (4):
  - Outeniqua Cancercare Oncology Unit, George, Eastern Cape
  - Cancercare Langenhoven, Port Elizabeth, Eastern Cape
  - Albert Alberts Stem Cell Transplant Research Centre, Pretoria, Gauteng
  - Constantiaberg Medi Clinic, Cape Town, Western Cape
- South Korea (4):
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Institut Català d'Oncologia Badalona, Badalona, Barcelona
  - Institut Català d'Oncologia Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Clinica Puerta de Hierro, Majadahonda, Madrid
  - Hospital Regional de Malaga | Oncologia, Málaga, Málaga
  - Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (2):
  - Phramongkutklao Hospital, Bangkok
  - Siriraj Hospital, Mahidol, Bangkok
- Turkey (Türkiye) (9):
  - Ankara Universitesi Tip Fakultesi Hastanesi, Ankara
  - Trakya Univ. Tip Fak., Edirne
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Marmara Uni. Tip Fak. Pendik EAH Hematoloji BD, Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
  - Ege Universitesi Tip Fakultesi, Izmir
  - Erciyes Universitesi Tip Fakultesi, Kayseri
  - Ondokuz Mayis Uni Tip Fakultesi, Samsun
  - Karadeniz Teknik Universitesi Tip Fakultesi, Trabzon
- Ukraine (5):
  - CNE "Clinical Center of Oncology, Hematology, Transplantology and Palliative Care of the Cherkasy Regional Council", Cherkasy
  - Municipal Non-Profit Enterprise "City Clinical Hospital ?4" of the Dnipro City Council, Dnipro
  - Clinic of National cancer institute - scientific and research department of pediatric oncology, Kyiv
  - State Institution - Institute of Blood Pathology and Transfusion Medicine NAMS of Ukraine, Lviv
  - CNE "Zaporizhzhia Regional Clinical Hospital" of Zaporizhzhia regional council, Zaporizhzhya
- United Kingdom (6):
  - Royal Devon & Exeter Hospital, Exeter, Devon
  - Northwick Park Hospital, Harrow, London
  - St George's Hospital, Kogarah, London
  - Dorset County Hospital, Dorchester
  - Royal Marsden Hospital (London), London
  - Singleton Hospital, Swansea

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Zinzani PL, Wang H, Feng J, Kim TM, Tao R, Zhang H, Fogliatto L, Maluquer Artigal C, Ozcan M, Yanez E, Kim WS, Kirtbaya D, Kriachok I, Maciel F, Xue H, Bouabdallah K, Phelps C, Chaturvedi S, Weispfenning A, Morcos PN, Odongo F, Buvaylo V, Childs BH, Dreyling M, Matasar M, Ghione P. CHRONOS-4: phase 3 study of copanlisib plus rituximab-based immunochemotherapy in relapsed indolent B-cell lymphoma. Blood Adv. 2024 Sep 24;8(18):4866-4876. doi: 10.1182/bloodadvances.2024013236. PMID 39058951
- [Derived] Matasar MJ, Dreyling M, Leppa S, Santoro A, Pedersen M, Buvaylo V, Fletcher M, Childs BH, Zinzani PL. Feasibility of Combining the Phosphatidylinositol 3-Kinase Inhibitor Copanlisib With Rituximab-Based Immunochemotherapy in Patients With Relapsed Indolent B-cell Lymphoma. Clin Lymphoma Myeloma Leuk. 2021 Nov;21(11):e886-e894. doi: 10.1016/j.clml.2021.06.021. Epub 2021 Jul 2. PMID 34389273
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: SRI part screened 42 participants from 12 countries, between 06-Jan-2016 (first participants first visit [FPFV]) and 31-Oct-2019 (last participant first visit [LPFV]). Phase 3 part screened 672 participants from 35 countries/regions, between 06-Feb-2017 (FPFV) and 31-Mar-2020(LPFV). Study terminated on 10-Nov-2023,
Pre-assignment Details: SRI: 42 participants were screened, 15 participants discontinued screening, 27 participants were enrolled and administered treatment. Phase 3: 672 participants were screened, 148 discontinued screening. 524 participants were enrolled and randomized to treatment. 4 participants were randomized but never administered, 520 participants were randomized and administered treatment.
Groups:
- SRI: Copa+R-B 45 mg: In SRI part, participants received copanlisib at dose level of 45 mg in combination with R-B.
- SRI: Copa+R-B 60 mg (Excluding Subjects From Japan): In SRI part, participants received copanlisib at dose level of 60 mg in combination with R-B.
- SRI: Copa+R-CHOP 45 mg: In SRI part, participants received copanlisib at dose level of 45 mg in combination with R-CHOP.
- SRI: Copa+R-CHOP 60 mg: In SRI part, participants received copanlisib at dose level of 60 mg in combination with R-CHOP.
- SRI: Japan Copa+R-B 60 mg: In SRI part, participants from Japan received copanlisib at dose level of 60 mg in combination with R-B.
- Phase 3: Copa+R-B/R-CHOP: In Phase 3 part, participants who never received R-B as a previous line of therapy were randomized to copanlisib + R-B. Participants who received R-B as a previous line of therapy were randomized to copanlisib + R-CHOP or, if progression-free interval after the last R-B treatment was ≥ 24 months, to copanlisib + R-B.
- Phase 3: Pbo+R-B/R-CHOP: In Phase 3 part, participants who never received R-B as a previous line of therapy were randomized to placebo + R-B. Participants who received R-B as a previous line of therapy were randomized to placebo + R-CHOP or, if progression-free interval after the last R-B treatment was ≥ 24 months, to placebo + R-B.
Period: Overall Study
Arm/Group | SRI: Copa+R-B 45 mg | SRI: Copa+R-B 60 mg (Excluding Subjects From Japan) | SRI: Copa+R-CHOP 45 mg | SRI: Copa+R-CHOP 60 mg | SRI: Japan Copa+R-B 60 mg | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Started | 3 | 7 | 5 | 6 | 6 | 262 | 262
Completed | 0 | 2 | 3 | 2 | 3 | 108 | 153
Not Completed | 3 | 5 | 2 | 4 | 3 | 154 | 109
Not completed — Other | 1 | 1 | 0 | 0 | 0 | 17 | 23
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 10 | 6
Not completed — Physician Decision | 0 | 2 | 2 | 2 | 1 | 10 | 3
Not completed — Patient decision: COVID-19 pandemic related | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician decision: COVID-19 pandemic related | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Logistical reason: COVID-19 pandemic related | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Patient decision | 0 | 1 | 0 | 0 | 1 | 36 | 22
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive disease - radiological progression | 0 | 0 | 0 | 0 | 0 | 11 | 22
Not completed — Progressive disease - clinical progression | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — AE not associated with clinical disease progression | 1 | 1 | 0 | 2 | 1 | 65 | 21
Not completed — AE associated with clinical disease progression | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Study intervention never administered | 0 | 0 | 0 | 0 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: FAS
Groups:
- Total: Total of all reporting groups
Arm/Group | SRI: Copa+R-B 45 mg | SRI: Copa+R-B 60 mg (Excluding Subjects From Japan) | SRI: Copa+R-CHOP 45 mg | SRI: Copa+R-CHOP 60 mg | SRI: Japan Copa+R-B 60 mg | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP | Total
Number analyzed (Participants) | 3 | 7 | 5 | 6 | 6 | 262 | 262 | 551
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 4 | 2 | 6 | 160 | 162 | 340
  >=65 years | 1 | 3 | 1 | 4 | 0 | 102 | 100 | 211
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 | 1 | 2 | 103 | 128 | 246
  Male | 0 | 2 | 1 | 5 | 4 | 159 | 134 | 305
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 24 | 32 | 56
  Not Hispanic or Latino | 3 | 7 | 5 | 5 | 6 | 223 | 215 | 464
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 15 | 15 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 2 | 0 | 0 | 6 | 98 | 82 | 189
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 4 | 1 | 6
  White | 2 | 5 | 3 | 6 | 0 | 144 | 168 | 328
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 15 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: SRI: Occurrence of Dose-limiting Toxicities (DLT)
Description: Dose-limiting toxicity is defined as any of the following occurring during Cycle 1 at a given dose level and regarded by the investigator and/or the sponsor to be possibly, probably, or definitely related to copanlisib given in combination with R-B or R-CHOP. General: any grade 5 hematologic or non-hematologic toxicity or any delay of >2 weeks of Cycle 2 due to study treatment-related toxicity; Non-hematologic DLT: any non-hematologic toxicity grade ≥ 3; Hematologic DLT: grade 4 absolute neutrophil count decrease lasting >7 days, or grade 4 febrile neutropenia, or grade 4 platelet count decreased or grade 3 platelet count decreased with serious bleeding, or signs of serious bleeding and/or international normalized ratio (INR) increased or partial thromboplastin time (PTT) prolonged of grade 3.
Time Frame: At Cycle 1: 28 days for Copa+R-B or 21 days for Copa+R-CHOP
Measure: Number; unit: Percentage
Arm/Group | SRI: Copa+R-B 45 mg | SRI: Copa+R-B 60 mg (Excluding Subjects From Japan) | SRI: Copa+R-CHOP 45 mg | SRI: Copa+R-CHOP 60 mg | SRI: Japan Copa+R-B 60 mg
Number analyzed (Participants) | 3 | 7 | 5 | 6 | 6
Percentage | 0 | 0 | 0 | 0 | 16.7

2. Primary Outcome: Phase 3: Progression-free Survival (PFS) by Independent Central Review
Description: PFS is defined as the time from randomization to progressive disease (PD) or death from any cause (if no progression is documented).
Time Frame: Approximately 6 years 4 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 262 | 262
Months | 32.9 [24.4 to 38.6] | 33.3 [27.8 to 42.8]
Statistical Analysis 1: Comparison: Phase 3: Copa+R-B/R-CHOP vs Phase 3: Pbo+R-B/R-CHOP; Test type: Superiority — Comparison of PFS; p = 0.827974, Log Rank — Significance level is 0.025; PFS was evaluated with a one-sided stratified log- rank test. HR and 95% CI are based on the stratified Cox regression model; Hazard Ratio (HR) = 1.125, 95% CI 2-sided [0.881 to 1.437]

3. Secondary Outcome: SRI: Best Overall Response
Description: Best overall response is defined as the best response achieved during the treatment and active follow-up periods; prior to end of study or start of new anti-tumor treatment, whichever occurs first.
Time Frame: Approximately 7 years 8 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | SRI: Copa+R-B 45 mg | SRI: Copa+R-B 60 mg (Excluding Subjects From Japan) | SRI: Copa+R-CHOP 45 mg | SRI: Copa+R-CHOP 60 mg | SRI: Japan Copa+R-B 60 mg
Number analyzed (Participants) | 3 | 7 | 5 | 6 | 6
Percentage
  Best response (BR) -Complete response (CR) | 33.3 (0.8) [0.8 to 90.6] | 71.4 (29.0) [29.0 to 96.3] | 60.0 (14.7) [14.7 to 94.7] | 16.7 (0.4) [0.4 to 64.1] | 50.0 (11.8) [11.8 to 88.2]
  BR - Very good partial response (VGPR) | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0]
  BR - Partial response (PR) | 66.7 (9.4) [9.4 to 99.2] | 28.6 (3.7) [3.7 to 71.0] | 20.0 (0.5) [0.5 to 71.6] | 83.3 (35.9) [35.9 to 99.6] | 33.3 (4.3) [4.3 to 77.7]
  BR - Minor response (MR) | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0]
  BR - Stable disease | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 20.0 (0.5) [0.5 to 71.6] | 0 (0) [0 to 0] | 0 (0) [0 to 0]
  BR - Progressive disease (PD) | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0]
  BR - Unconfirmed early stable disease (uSD) | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0]
  BR - Not evaluable | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 16.7 (0.4) [0.4 to 64.1]
  BR - Not available | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0]
  Response rate - Objective response rate (ORR) | 100.0 (29.2) [29.2 to 100.0] | 100.0 (59.0) [59.0 to 100.0] | 80.0 (28.4) [28.4 to 99.5] | 100.0 (54.1) [54.1 to 100.0] | 83.3 (35.9) [35.9 to 99.6]
  Response rate - Disease control rate (DCR) | 100.0 (29.2) [29.2 to 100.0] | 100.0 (59.0) [59.0 to 100.0] | 100.0 (47.8) [47.8 to 100.0] | 100.0 (54.1) [54.1 to 100.0] | 83.3 (35.9) [35.9 to 99.6]
  Response rate - Complete response rate (CRR) | 33.3 (0.8) [0.8 to 90.6] | 71.4 (29.0) [29.0 to 96.3] | 60.0 (14.7) [14.7 to 94.7] | 16.7 (0.4) [0.4 to 64.1] | 50.0 (11.8) [11.8 to 88.2]

4. Secondary Outcome: SRI: Number of Subjects With Treatment-emergent Adverse Event (TEAE)
Description: A treatment-emergent AE is defined as any event arising or worsening after start of study drug administration until 30 days after the last study drug intake.
Time Frame: Approximately 4 years 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | SRI: Copa+R-B 45 mg | SRI: Copa+R-B 60 mg (Excluding Subjects From Japan) | SRI: Copa+R-CHOP 45 mg | SRI: Copa+R-CHOP 60 mg | SRI: Japan Copa+R-B 60 mg
Number analyzed (Participants) | 3 | 7 | 5 | 6 | 6
Participants
  Any TEAE | 3 | 7 | 5 | 6 | 6
  TESAEs | 2 | 3 | 3 | 6 | 3

5. Secondary Outcome: Phase 3: Objective Tumor Response Rate (ORR)-Independent Central Review
Description: ORR, as assessed by independent central review, is defined as the percentage of participants who had a best response rating of CR or PR according to the Lugano classification and for subjects with LPL/WM, a response rating of CR, VGPR, PR, or MR according to the Owen criteria, over the whole duration of the study (i.e., until time of analysis of PFS).
Time Frame: Up to 6 years 4 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 262 | 262
Percentage | 85.5 (80.6) [80.6 to 89.5] | 86.6 (81.9) [81.9 to 90.5]
Statistical Analysis 1: Comparison: Phase 3: Copa+R-B/R-CHOP vs Phase 3: Pbo+R-B/R-CHOP; Test type: Superiority — ORR of Copa+R-B/R-CHOP minus ORR of Pbo+R-B/R-CHOP; p = 0.658652, Cochran-Mantel-Haenszel — Significance level is 0.025. P-values are descriptive (nominal) due to multiplicity testing; Point estimate and 95% CI are based on Mantel-Haenszel weighted treatment difference; Difference = -1.25, 95% CI 2-sided [-7.25 to 4.75]

6. Secondary Outcome: Phase 3: ORR-Investigator Assessment
Description: ORR, as assessed by investigator, is defined as the percentage of participants who had a best response rating of CR or PR according to the Lugano classification and for subjects with LPL/WM, a response rating of CR, VGPR, PR, or MR according to the Owen criteria, over the whole duration of the study (i.e., until time of analysis of PFS).
Time Frame: Up to 6 years 4 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 262 | 262
Percentage | 85.5 (80.6) [80.6 to 89.5] | 86.6 (81.9) [81.9 to 90.5]
Statistical Analysis 1: Comparison: Phase 3: Copa+R-B/R-CHOP vs Phase 3: Pbo+R-B/R-CHOP; Test type: Superiority — ORR of Copa+R-B/R-CHOP minus ORR of Pbo+R-B/R-CHOP; p = 0.605183, Cochran-Mantel-Haenszel — Significance level is 0.025. P-value is descriptive (nominal) due to multiplicity testing; Point estimate and 95% CI are based on Mantel-Haenszel weighted treatment difference; Difference = -0.80, 95% CI 2-sided [-6.64 to 5.05]

7. Secondary Outcome: Phase 3: Duration of Tumor Response (DOR)-Independent Central Review
Description: DOR, as assessed by independent central review, is defined as the time (in days) from first observed tumor response (CR, VGPR, PR, or MR) until progression or death from any cause, whichever occurred earlier. The DOR was only defined for patients with at least 1 CR, VGPR, PR, or MR.
Time Frame: Approximately 6 years 4 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 224 | 227
Months | 32.2 (22.8) [22.8 to 38.8] | 32.4 (27.7) [27.7 to 42.0]
Statistical Analysis 1: Comparison: Phase 3: Copa+R-B/R-CHOP vs Phase 3: Pbo+R-B/R-CHOP; Test type: Superiority — Comparison of DOR; p = 0.846204, Log Rank — Significance level is 0.025, P-value is descriptive (nominal) due to multiplicity testing; DOR was evaluated with a one-sided stratified log-rank test. HR and its 95% CI were based on the stratified Cox regression model; Hazard Ratio (HR) = 1.145, 95% CI 2-sided [0.883 to 1.484]

8. Secondary Outcome: Phase 3: DOR-Investigator Assessment
Description: DOR, as assessed by investigator, is defined as the time (in days) from first observed tumor response (CR, VGPR, PR, or MR) until progression or death from any cause, whichever occurred earlier. The DOR was only defined for patients with at least 1 CR, VGPR, PR, or MR.
Time Frame: Approximately 6 years 4 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 227 | 229
Months | 32.4 [24.3 to 38.8] | 30.9 [24.8 to 42.0]
Statistical Analysis 1: Comparison: Phase 3: Copa+R-B/R-CHOP vs Phase 3: Pbo+R-B/R-CHOP; Test type: Superiority — Comparison of DOR; p = 0.801735, Log Rank — Significance level is 0.025, P-value is descriptive (nominal) due to multiplicity testing; [statistical method as in outcome 7, analysis 1]; Hazard Ratio (HR) = 1.117, 95% CI 2-sided [0.865 to 1.443]

9. Secondary Outcome: Phase 3: Complete Tumor Response Rate (CRR)-Independent Central Review
Description: CRR, as assessed by independent central review, is defined as the proportion of patients who had a best response rating of CR according to the Lugano classification, and for patients with LPL/WM, a response rating of CR according to the Owen criteria, over the whole duration of the study (i.e., until the time of analysis of PFS).
Time Frame: Approximately 6 years 4 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 262 | 262
Percentage | 38.5 (32.6) [32.6 to 44.7] | 41.2 (35.2) [35.2 to 47.4]
Statistical Analysis 1: Comparison: Phase 3: Copa+R-B/R-CHOP vs Phase 3: Pbo+R-B/R-CHOP; Test type: Superiority — CRR of Copa+R-B/R-CHOP minus CRR of Pbo+R-B/R-CHOP; p = 0.741153, Cochran-Mantel-Haenszel — Significance level is 0.025. P-value is descriptive (nominal) due to multiplicity testing; Point estimate and 95% CI are based on Mantel-Haenszel weighted treatment difference; Difference = -2.74, 95% CI 2-sided [-11.06 to 5.57]

10. Secondary Outcome: Phase 3: CRR-Investigator Assessment
Description: CRR, as assessed by investigator, is defined as the proportion of patients who had a best response rating of CR according to the Lugano classification, and for patients with LPL/WM, a response rating of CR according to the Owen criteria, over the whole duration of the study (i.e., until the time of analysis of PFS).
Time Frame: Approximately 6 years 4 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 262 | 262
Percentage | 39.7 [33.7 to 45.9] | 42.0 [35.9 to 48.2]
Statistical Analysis 1: Comparison: Phase 3: Copa+R-B/R-CHOP vs Phase 3: Pbo+R-B/R-CHOP; Test type: Superiority — CRR of Copa+R-B/R-CHOP minus CRR of Pbo+R-B/R-CHOP; p = 0.696482, Cochran-Mantel-Haenszel — Significance level is 0.025. P-value is descriptive (nominal) due to multiplicity testing; Point estimate and 95% CI are based on Mantel-Haenszel weighted treatment difference; Difference = -2.21, 95% CI 2-sided [-10.62 to 6.20]

11. Secondary Outcome: Phase 3: Disease Control Rate (DCR)-Independent Central Review
Description: DCR, as assessed by independent central review, is defined as the proportion of patients who had a best response rating of CR, VGPR, PR, MR, or stable disease (excluding unconfirmed early stable disease).
Time Frame: Approximately 6 years 4 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 262 | 262
Percentage | 88.5 (84.1) [84.1 to 92.1] | 92.4 (88.5) [88.5 to 95.3]
Statistical Analysis 1: Comparison: Phase 3: Copa+R-B/R-CHOP vs Phase 3: Pbo+R-B/R-CHOP; Test type: Superiority — DCR of Copa+R-B/R-CHOP minus DCR of Pbo+R-B/R-CHOP; p = 0.936009, Cochran-Mantel-Haenszel — Significance level is 0.025. P-value is descriptive (nominal) due to multiplicity testing; Point estimate and 95% CI are based on Mantel-Haenszel weighted treatment difference; Difference = -3.95, 95% CI 2-sided [-9.04 to 1.14]

12. Secondary Outcome: Phase 3: DCR-Investigator Assessment
Description: DCR, as assessed by investigator, is defined as the proportion of patients who had a best response rating of CR, VGPR, PR, MR, or stable disease (excluding unconfirmed early stable disease).
Time Frame: Approximately 6 years 4 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 262 | 262
Percentage | 88.5 (84.1) [84.1 to 92.1] | 92.4 (88.5) [88.5 to 95.3]
Statistical Analysis 1: Comparison: Phase 3: Copa+R-B/R-CHOP vs Phase 3: Pbo+R-B/R-CHOP; Test type: Superiority — DCR of Copa+R-B/R-CHOP minus DCR of Pbo+R-B/R-CHOP; p = 0.944242, Cochran-Mantel-Haenszel — Significance level is 0.025. P-value is descriptive (nominal) due to multiplicity testing; Point estimate and 95% CI are based on Mantel-Haenszel weighted treatment difference; Difference = -3.89, 95% CI 2-sided [-8.68 to 0.90]

13. Secondary Outcome: Phase 3: Time to Tumor Progression (TTP)-Independent Central Review
Description: TTP, as assessed by independent central review, is defined as the time from randomization to progression or death related to progression, whichever occurred earlier. Death related to progression was any death except for: death due to an AE unrelated to progression; or death with a specification of "other" as reason (which excludes PD).
Time Frame: Approximately 6 years 4 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 262 | 262
Months | 36.1 (30.3) [30.3 to 44.0] | 35.0 (30.4) [30.4 to 44.8]
Statistical Analysis 1: Comparison: Phase 3: Copa+R-B/R-CHOP vs Phase 3: Pbo+R-B/R-CHOP; Test type: Superiority — Comparison of TTP; p = 0.517849, Log Rank — Significance level is 0.025. P-value is descriptive (nominal) due to multiplicity testing; TTP was evaluated with a one-sided stratified log-rank test. HR and its 95% CI are based on the stratified Cox regression model; Hazard Ratio (HR) = 1.006, 95% CI 2-sided [0.777 to 1.303]

14. Secondary Outcome: Phase 3: TTP-Investigator Assessment
Description: TTP, as assessed by investigator, is defined as the time from randomization to progression or death related to progression, whichever occurred earlier. Death related to progression was any death except for: death due to an AE unrelated to progression; or death with a specification of "other" as reason (which excludes PD).
Time Frame: Approximately 6 years 4 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 262 | 262
Months | 36.1 (30.3) [30.3 to 44.0] | 35.0 (30.4) [30.4 to 44.8]
Statistical Analysis 1: Comparison: Phase 3: Copa+R-B/R-CHOP vs Phase 3: Pbo+R-B/R-CHOP; Test type: Superiority — Comparison of TTP; p = 0.411398, Log Rank — Significance level is 0.025. P-value is descriptive (nominal) due to multiplicity testing; [statistical method as in outcome 13, analysis 1]; Hazard Ratio (HR) = 0.971, 95% CI 2-sided [0.750 to 1.257]

15. Secondary Outcome: Phase 3: Time to Next Anti-lymphoma Treatment (TTNT)
Description: A new anti-lymphoma therapy is any new systemic anticancer treatment or radiotherapy for lymphoma, with a consolidation intent. TTNT was defined as the time from the date of randomization to the start of new anti-lymphoma therapy, where the date of randomization was considered Day 1.
Time Frame: Approximately 6 years 4 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 262 | 262
Months | NA [50.1 to NA] — NA: Value cannot be estimated due to censored data, insufficient number of participants with events. | NA [NA to NA] — NA: Value cannot be estimated due to censored data, insufficient number of participants with events.
Statistical Analysis 1: Comparison: Phase 3: Copa+R-B/R-CHOP vs Phase 3: Pbo+R-B/R-CHOP; Test type: Superiority — Comparison of TTNT; p = 0.955865, Log Rank — Significance level IS 0.025. P-value is descriptive (nominal) due to multiplicity testing; TTNT was evaluated with a one-sided stratified log-rank test. HR and its 95% CI are based on the stratified Cox regression model; Hazard Ratio (HR) = 1.289, 95% CI 2-sided [0.962 to 1.728]

16. Secondary Outcome: Phase 3: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization until death from any cause. The OS for patients alive at the time of the database cut-off date was censored to the last date they were known to be alive. Deaths that occurred after the database cut-off date, reported during data cleaning, were considered for establishing the last known alive date at data cut-off.
Time Frame: Approximately 6 years 4 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 262 | 262
Months | NA [NA to NA] — NA: Value cannot be estimated due to censored data, insufficient number of participants with events. | NA [NA to NA] — NA: Value cannot be estimated due to censored data, insufficient number of participants with events.
Statistical Analysis 1: Comparison: Phase 3: Copa+R-B/R-CHOP vs Phase 3: Pbo+R-B/R-CHOP; Test type: Superiority — Comparison of OS; p = 0.758563, Log Rank — Significance level is 0.025. P-value is descriptive (nominal) due to multiplicity testing; OS was evaluated with a one-sided stratified log-rank test. HR and 95% CI are based on the stratified Cox regression model; Hazard Ratio (HR) = 1.132, 95% CI 2-sided [0.800 to 1.603]

17. Secondary Outcome: Phase 3: Time to Deterioration in Disease-related Symptoms-physical (DRS-P) of at Least 3 Points of Lymphoma
Description: Time to deterioration in DRS-P of at least 3 points, as measured by the FLymSI-18 questionnaire, was evaluated in all patients. It is defined as the time from randomization to DRS-P decline, progression, or death from any reason, whichever occurred earlier.
Time Frame: Approximately 6 years 4 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 262 | 262
Months | 2.7 (1.9) [1.9 to 3.3] | 6.3 (4.6) [4.6 to 8.3]
Statistical Analysis 1: Comparison: Phase 3: Copa+R-B/R-CHOP vs Phase 3: Pbo+R-B/R-CHOP; Test type: Superiority — Comparison of time to deterioration in DRS-P; p = 0.999695, Log Rank — Significance level IS 0.025. P-value is descriptive (nominal) due to multiplicity testing; Time to deterioration in DRS-P was evaluated with one-sided stratified log-rank test.HR and its 95% CI are based on stratified Cox regression model; Hazard Ratio (HR) = 1.394, 95% CI 2-sided [1.149 to 1.691]

18. Secondary Outcome: Phase 3: Time to Improvement in Disease-related Symptoms-physical (DRS-P) of at Least 3 Points of Lymphoma
Description: Time to improvement in DRS-P of at least 3 points, as measured by the FLymSI-18 questionnaire, was evaluated for all patients. It is defined as the time from randomization to DRS-P improvement of at least 3 points.
Time Frame: Approximately 6 years 4 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 262 | 262
Months | 12.8 (6.7) [6.7 to 36.1] | 5.1 (2.8) [2.8 to 8.3]
Statistical Analysis 1: Comparison: Phase 3: Copa+R-B/R-CHOP vs Phase 3: Pbo+R-B/R-CHOP; Test type: Superiority — Comparison of time to improvement in DRS-P; p = 0.965639, Log Rank — Significance level is 0.025. P-value is descriptive (nominal) due to multiplicity testing; Time to improvement in DRS-P was evaluated with one-sided stratified log-rank test.HR and its 95% CI are based on the stratified Cox regression model; Hazard Ratio (HR) = 0.810, 95% CI 2-sided [0.642 to 1.020]

19. Secondary Outcome: Phase 3: Number of Subjects With Treatment-emergent Adverse Event (TEAE)
Description: as for outcome 4
Time Frame: Approximately 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
Number analyzed (Participants) | 263 | 257
Participants
  Any TEAE | 263 | 250
  TESAEs | 161 | 54
  Any copanlisib or placebo related TEAE | 250 | 214
  Any copanlisib or placebo related TESAEs | 118 | 26
  Any R-B/R-CHOP related TEAE | 245 | 224
  Any R-B/R-CHOP related TESAEs | 109 | 26

ADVERSE EVENTS:
Time Frame: After the first study intervention up to 30 days after the end of study intervention. For SRI, this is over a period of approximately 4 years 10 months and for phase 3, over a period of approximately 4 years.
Description: Adverse event reporting, for the all-cause mortality, considers all deaths that occurred at any time during the study before the last contact. For SRI, up to 7 years 8 months. For phase 3, up to 6 years 4 months.
Groups:
- SRI: Copa+R-B 45 mg: In SRI part, subjects received 45 mg of copanlisib in combination with R-B.
- SRI: Copa+R-B 60 mg (Excluding Subjects From Japan): In SRI part, subjects received 60 mg of copanlisib in combination with R-B.
- SRI: Copa+R-CHOP 45 mg: In SRI part, subjects received 45 mg of copanlisib in combination with R-CHOP.
- SRI: Copa+R-CHOP 60 mg: In SRI part, subjects received 60 mg of copanlisib in combination with R-CHOP.
- SRI: Japan Copa+R-B 60 mg: In SRI part, Subjects from Japan only received 60 mg of copanlisib in combination with R-B.
Arm/Group | SRI: Copa+R-B 45 mg | SRI: Copa+R-B 60 mg (Excluding Subjects From Japan) | SRI: Copa+R-CHOP 45 mg | SRI: Copa+R-CHOP 60 mg | SRI: Japan Copa+R-B 60 mg | Phase 3: Copa+R-B/R-CHOP | Phase 3: Pbo+R-B/R-CHOP
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/7 | 0/5 | 1/6 | 0/6 | 68/263 | 62/257
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/7 | 3/5 | 6/6 | 3/6 | 161/263 | 54/257
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 5/5 | 6/6 | 6/6 | 259/263 | 250/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SRI: Copa+R-B 45 mg (N=3) | SRI: Copa+R-B 60 mg (Excluding Subjects From Japan) (N=7) | SRI: Copa+R-CHOP 45 mg (N=5) | SRI: Copa+R-CHOP 60 mg (N=6) | SRI: Japan Copa+R-B 60 mg (N=6) | Phase 3: Copa+R-B/R-CHOP (N=263) | Phase 3: Pbo+R-B/R-CHOP (N=257)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (4)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 18 (18) | 8 (8)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 5 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 1 (1) | 22 (26) | 4 (5)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related hypersensitivity reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (16) | 2 (2)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disseminated cryptococcosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 34 (38) | 3 (3)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (2)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ludwig angina (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective thrombosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (8) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Cytomegalovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Norovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 10 (11) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SRI: Copa+R-B 45 mg (N=3) | SRI: Copa+R-B 60 mg (Excluding Subjects From Japan) (N=7) | SRI: Copa+R-CHOP 45 mg (N=5) | SRI: Copa+R-CHOP 60 mg (N=6) | SRI: Japan Copa+R-B 60 mg (N=6) | Phase 3: Copa+R-B/R-CHOP (N=263) | Phase 3: Pbo+R-B/R-CHOP (N=257)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (10) | 2 (3) | 3 (5) | 0 (0) | 85 (166) | 64 (147)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 3 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 8 (11) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (8) | 1 (1) | 0 (0) | 0 (0) | 13 (18) | 21 (39)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 15 (29) | 22 (42)
Neutropenia (Blood and lymphatic system disorders) | 2 (5) | 5 (24) | 4 (20) | 1 (1) | 1 (1) | 86 (213) | 88 (232)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 3 (7) | 2 (8) | 1 (3) | 0 (0) | 44 (68) | 28 (57)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 14 (17) | 14 (17)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 12 (13) | 13 (14)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (4) | 3 (5) | 1 (1) | 0 (0) | 36 (43) | 49 (57)
Diarrhoea (Gastrointestinal disorders) | 1 (4) | 3 (5) | 3 (5) | 4 (4) | 2 (4) | 88 (137) | 38 (45)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (11) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (10) | 8 (13)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 8 (8) | 7 (7)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 16 (21) | 4 (5)
Nausea (Gastrointestinal disorders) | 3 (6) | 5 (8) | 3 (3) | 1 (1) | 4 (4) | 112 (208) | 92 (156)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 4 (5) | 0 (0) | 2 (2) | 1 (4) | 25 (31) | 10 (10)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 59 (123) | 31 (44)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (6) | 1 (1) | 0 (0) | 0 (0) | 18 (20) | 21 (28)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 18 (24) | 6 (9)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Fatigue (General disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 51 (65) | 49 (63)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 26 (47) | 15 (26)
Mucosal inflammation (General disorders) | 1 (1) | 1 (6) | 0 (0) | 1 (1) | 0 (0) | 9 (14) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 4 (6) | 2 (2) | 2 (2) | 2 (4) | 87 (130) | 34 (51)
Swelling face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 14 (16) | 7 (10)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 5 (5)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 47 (70) | 14 (14)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 13 (14) | 15 (16)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (10) | 5 (7)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 14 (16) | 11 (15)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 9 (9) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 10 (12) | 7 (7)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 31 (34) | 4 (4)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 5 (5) | 9 (10)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 3 (4) | 44 (63) | 37 (51)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 19 (32) | 17 (22)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 14 (29) | 4 (6)
Borrelia infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 8 (10) | 4 (7)
Erythema migrans (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 9 (13) | 15 (17)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 38 (62) | 22 (38)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 13 (15) | 10 (17)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 3 (4) | 34 (51) | 18 (27)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 19 (33) | 13 (27)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 12 (23) | 7 (8)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 9 (11) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 9 (11) | 14 (17)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 27 (53) | 11 (14)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 8 (13) | 3 (3)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 16 (16) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 6 (7)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 15 (16) | 7 (9)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 18 (21) | 13 (18)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (6) | 72 (232) | 50 (145)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 2 (6) | 3 (5) | 109 (489) | 82 (301)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (5) | 3 (3) | 1 (1) | 72 (209) | 52 (126)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 64 (74) | 21 (29)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (6) | 78 (386) | 65 (272)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Cytomegalovirus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 20 (28) | 13 (22)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 20 (28) | 7 (11)
Inflammatory marker increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudomonas test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Norovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 6 (15) | 5 (8) | 3 (3) | 4 (4) | 150 (318) | 53 (145)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 26 (40) | 17 (24)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 21 (34)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 13 (16) | 2 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 11 (16) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 44 (62) | 9 (13)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 24 (29) | 8 (10)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 1 (2) | 43 (54) | 32 (40)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 8 (11) | 15 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 11 (12) | 23 (31)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 3 (3)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 8 (8) | 7 (7)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 18 (22) | 12 (17)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 9 (21) | 10 (11)
Headache (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 35 (44) | 29 (42)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 4 (5)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 3 (3)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Vagus nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 23 (29) | 13 (13)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (5)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 3 (3)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 41 (59) | 37 (47)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 14 (15) | 11 (12)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 9 (10) | 7 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (12) | 10 (10)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 6 (14) | 3 (3)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 6 (6)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 30 (39) | 24 (29)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (8) | 0 (0) | 1 (1) | 1 (1) | 59 (75) | 26 (33)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 25 (38) | 14 (16)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (3)
Ureteral stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (10) | 4 (6) | 3 (3) | 3 (3) | 114 (328) | 42 (90)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 8 (18) | 7 (9)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 11 (12) | 6 (6)
Secondary hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT02626455/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT02626455/SAP_001.pdf